CLINICAL TRIAL: NCT01656733
Title: Nicotine Replacement for Smoking Cessation During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Cheryl Oncken, Professor of Medicine, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-057-6; 1R01HD069314-01A1 (NIH)
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Nicotine Dependence; Smoking Cessation
Keywords: Smoking Cessation; Pregnancy; Nicotrol Inhaler; Placebo Inhaler; Nicotine Inhaler
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotrol Inhaler (Experimental): Nicotrol Inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper.
  Interventions: Drug: Nicotrol Inhaler
- Placebo Inhaler (Placebo Comparator): Placebo inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper
  Interventions: Drug: Placebo Inhaler

INTERVENTIONS:
Drug: Nicotrol Inhaler — Nicotrol Inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper
  Other Names: Nicotine Inhaler
  Arms: Nicotrol Inhaler
Drug: Placebo Inhaler — Placebo inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper
  Arms: Placebo Inhaler

SUMMARY:
This is a clinical trial to determine if the nicotine inhaler in combination with counseling will help pregnant women quit smoking, and whether it is safe when compared to placebo (an inactive inhaler).

DETAILED DESCRIPTION:
This project will examine the safety and efficacy of the nicotine inhaler as an aid to smoking cessation during pregnancy. The specific aims are: (1) To examine the efficacy of the nicotine inhaler compared to a matching placebo for smoking cessation during pregnancy; (2) To compare the nicotine inhaler with placebo on overall nicotine exposure (i.e., serum cotinine concentrations), and on birth outcomes (i.e., birth weight and gestational age); (3) To identify factors that determine which women benefit most from the use of the nicotine inhaler for smoking cessation during pregnancy; (4) To explore mechanisms by which the nicotine inhaler increases birth weight and gestational age.

Subjects will be recruited from two prenatal clinics that serve primarily a low-income, minority population.

Pregnant smokers (n=270) who smoke at least 5 cigarettes/ day will receive nurse-delivered behavioral counseling and be randomized to receive a 6-week course of treatment with either a nicotine inhaler or placebo, followed by a 6-week taper. Birth outcomes will be obtained on all participants

ELIGIBILITY:
Inclusion Criteria:

* smoking at least 5 cigarettes per day for the preceding 7 days
* previous attempt to quit smoking during pregnancy by self report
* 13-26 weeks gestation
* at least 16 years of age
* able to speak English or Spanish
* intent to carry pregnancy to term
* stable residence

Exclusion Criteria:

* current drug or alcohol abuse or dependence (other than methadone maintenance)
* twins or other multiple gestation
* unstable psychiatric disorder
* unstable medical problems (e.g., pre-eclampsia, threatened abortion, hyperemesis gravidarum)
* known congenital abnormality

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-08; Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Oncken, M.D., M.P.H., Principal Investigator — UConn Health
Locations (2):
- United States (2):
  - Women's Ambulatory Health Services at Hartford Hospital, Hartford, Connecticut
  - Wesson Women's Clinic at Baystate Medical Center, Springfield, Massachusetts

REFERENCES:
- [Derived] Oncken C, Dornelas EA, Kuo CL, Sankey HZ, Kranzler HR, Mead EL, Thurlow MSD. Randomized Trial of Nicotine Inhaler for Pregnant Smokers. Am J Obstet Gynecol MFM. 2019 Mar;1(1):10-18. doi: 10.1016/j.ajogmf.2019.03.006. Epub 2019 Mar 27. PMID 31380506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited beginning August 20, 2012. Enrollment sites included Hartford Hospital (Hartford, CT) and Baystate Medical Center (Springfield, MA).
Pre-assignment Details: 154 participants gave written consent for study participation and 137 were randomized. Therefore, 17 participants were excluded for the following reasons: no show after screen (10), high PHQ9 (2), moved out of area (2), current drug use (1), advanced gestational age (1), and stress too high to continue (1).
Groups:
- Placebo Inhaler: Placebo inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper
  Nicotrol Inhaler: Nicotrol Inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper Placebo Inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper.
- Nicotrol Inhaler: Nicotrol Inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper.
  Nicotrol Inhaler: Nicotrol Inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper Placebo Inhaler, 1-12 cartridges per day, for 6 weeks with a 6 week taper.
Period: Overall Study
Arm/Group | Placebo Inhaler | Nicotrol Inhaler
Started (Baseline Visit (randomization)) | 67 (4 discontinued after BL visit (lost to follow up)) | 70 (5 discontinued after BL visit ( lost to follow up))
Visit 1 (1 Week After Quit Date) | 45 | 42
Visit 2 (2 Weeks After Quit Date) | 32 | 44
Visit 3 (3 Weeks After Quit Date) | 33 | 34
Visit 4 (4 Weeks After Quit Date) | 32 | 30
Visit 5 (6 Weeks After Quit Date) | 37 | 36
Visit 6 ( 32-36 Weeks Gestation) | 39 | 47
Participants With Perinatal Outcomes | 67 | 66
Visit 7 (1 Month Postpartum) Phone Call | 47 | 50
Visit 8 (6 Months Postpartum) | 30 | 28
Completed | 67 | 66
Not Completed | 0 | 4
Not completed — No permission to collect birth outcomes | 0 | 1
Not completed — Delivery at another hospital | 0 | 2
Not completed — Spontaneous abortion | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Inhaler | Nicotrol Inhaler | Total
Number analyzed (Participants) | 67 | 70 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.24 (6.30) | 26.97 (5.45) | 27.59 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 70 | 137
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 28 | 61
  Non-Hispanic, White | 25 | 26 | 51
  Non-Hispanic, Black | 8 | 14 | 22
  Other | 0 | 1 | 1
  Unknown | 1 | 1 | 2
Highest level of education completed [Number; unit: participants]
  Grade School Completed | 20 | 18 | 38
  High School Completed | 31 | 36 | 67
  College or post college completed | 16 | 16 | 32
Number of Cigs/day [Mean (Standard Deviation); unit: cigarettes per day] — number of cigarettes per day reported at baseline
  cigarettes per day | 8.04 (4.59) | 8.66 (4.71) | 8.36 (4.64)
Number of cigarettes per day last two weeks [Mean (Standard Deviation); unit: cigarettes per day] | 5.03 (4.69) | 3.48 (3.29) | 4.14 (3.99)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self Report an Average of Zero Cigarettes Smoked Per Day in Preceding 7 Days
Description: Number of participants who self report an average of zero cigarettes smoked per day in preceding 7 days
Time Frame: 32-34 weeks gestation (Visit 6)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Inhaler | Nicotrol Inhaler
Number analyzed (Participants) | 67 | 70
Participants | 12 | 7

2. Secondary Outcome: Exhaled Carbon Monoxide
Description: As measured by parts per million (ppm) on CO breathalyzer
Time Frame: 32-34 weeks gestation
Population: Overall number of participants includes only those that attended the 32-34 gestation week visit
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Placebo Inhaler | Nicotrol Inhaler
Number analyzed (Participants) | 40 | 46
parts per million | 5.50 (5.42) | 6.7 (7.4)

3. Secondary Outcome: Birth Weight
Description: Birth weight in grams
Time Frame: At delivery
Population: Could not obtain birth outcomes on 4 individuals in nicotine group for various reasons.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Placebo Inhaler | Nicotrol Inhaler
Number analyzed (Participants) | 67 | 66
Grams | 3036.78 (583.8) | 3141.12 (561.94)

4. Secondary Outcome: Gestational Age
Description: Measure of age of pregnancy at delivery
Time Frame: At delivery
Population: Could not obtain birth outcomes on 4 individuals in nicotine group for various reasons.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Placebo Inhaler | Nicotrol Inhaler
Number analyzed (Participants) | 67 | 66
weeks | 38.61 (2.53) | 39.11 (2.42)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline visit up to delivery of infant.
Arm/Group | Placebo Inhaler | Nicotrol Inhaler
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/70
Serious Adverse Events (participants affected / at risk) | 40/67 | 28/70
Other Adverse Events (participants affected / at risk) | 0/67 | 12/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Inhaler (N=67) | Nicotrol Inhaler (N=70)
Low Birth Weigh (<2500 grams) (Pregnancy, puerperium and perinatal conditions) | 10 | 4
Preterm delivery (Pregnancy, puerperium and perinatal conditions) | 10 | 3
Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Perinatal Mortality (Pregnancy, puerperium and perinatal conditions) | 0 | 0
Neonatal Abstinence Syndrome (Pregnancy, puerperium and perinatal conditions) | 11 | 13
Maternal Hospitalizationfor Medical Condition (Pregnancy, puerperium and perinatal conditions) | 1 | 3
Fetal Cardiac Anomaly (Cardiac disorders) | 1 | 0
Right Club Foot (Congenital, familial and genetic disorders) | 1 | 0
Infant Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Infant Low Blood Sugar (Endocrine disorders) | 1 | 1
Infant Bradycardia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Inhaler (N=67) | Nicotrol Inhaler (N=70)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Bad taste (General disorders) | 0 | 1
Increased mucus in throat (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT01656733/Prot_SAP_000.pdf